CLINICAL TRIAL: NCT03552887
Title: Adverse Events During Physiotherapy at Intensive Care Unit In Patients Undergoing Cardiac Surgery
Acronym: Adephysio
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Emilia Nozawa, PT PhD, Vice Director, Physiotherapy Department, University of Sao Paulo General Hospital
Other Study IDs: 1391854; 51256215.5.0000.0068 (Other: CAAE)
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Adverse Event; Physiotherapy; Intensive Care Units; Cardiac Surgery; Postoperative
Keywords: Adverse Event; Physiotherapy; Cardiac Surgery
MeSH Terms: interventions — Cardiac Surgical Procedures; Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postoperative patients: Cohort of patients undergoing cardiac surgery, aged ≥ 18 years old, who had received any physiotherapy intervention
  Interventions: Procedure: Cardiac Surgery; Procedure: Physiotherapy

INTERVENTIONS:
Procedure: Cardiac Surgery — Any type of cardiac surgery
Procedure: Physiotherapy — Any type of physiotherapy intervention, performed by physiotherapists outside of the protocol

SUMMARY:
This study aims to estimate the incidence of adverse events during physiotherapy at intensive care unit (ICU) in adult patients undergoing cardiac surgery and to identify predictors of those events. This is a prospective cohort study, and the investigators observed all types of physiotherapy interventions in patients admitted at surgical ICU.

DETAILED DESCRIPTION:
Physiotherapy intervention practice in patients after cardiac surgery has been associated with better clinical outcomes, but the safety of such interventions are not fully understood.

A prospective observational study of patients admitted at surgical ICU, aged > 18 years old, undergoing cardiac surgery was conducted to estimate the incidence of adverse events during physiotherapy interventions in those patients and to identify predictors of adverse events.

Physiotherapy interventions were observed, performed by physiotherapists outside of the protocol. The occurrence of adverse events or physiological abnormality were recorded, classifying them according to the symptomatic consequences for the patient, from grade 1 ("near miss", additional intervention not required) to grade 5 (death). The investigators collected clinical characteristics of patients, such as sequential organ failure assessment (SOFA) score, comorbidities, sedation leve and pain. Participants were followed up to hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery
* Age ≥ 18 years old
* Patients who are receiving any physiotherapy intervention

Exclusion Criteria:

* Neurological and cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted at surgical ICU, undergoing cardiac surgery, and who had receive any physiotherapy intervention, at Instituto do Coracao - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, Brazil
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Adverse Event | until date of ICU discharge or date of death from any cause, whichever came first, up to 24 months
  Occurrence of adverse events during all physiotherapy interventions.

SECONDARY OUTCOMES:
Grade of adverse event | until date of ICU discharge or date of death from any cause, whichever came first, up to 24 months
  Grade of observed adverse event according to the symptomatic consequences for the patient, from grade 1 ("near miss", additional intervention not required) to grade 5 (death)
Mortality Rate | Until hospital discharge, up to 24 months
  Number of deaths
ICU Length of Stay | Until ICU discharge, up to 24 months
  Number of days in ICU
Hospital Length of Stay | Until hospital discharge, up to 24 months
  Number of days in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Nozawa, PhD, PT, Principal Investigator — Instituto do Coracao, Hospital das Clinicas, USP

IPD SHARING:
Plan to Share IPD: No
No individual personal data will be disclosed